CLINICAL TRIAL: NCT02633072
Title: Evaluation of the Visual Acuity After the Implantation of a Tecnis +2.75 Diopters Bifocal Intraocular Lens (Tecnis ZKB00) in the Distance Dominant Eye, in Combination With a +3.25 Diopters Tecnis Bifocal Intraocular Lens (Tecnis ZLB00) in the Fellow Eye.
Brief Title: Visual Acuity After the Combined Binocular Implantation of +2.75 Diopters and +3.25 Diopters Tecnis Multifocal Intraocular Lenses.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PD Dr. med. Eckart Bertelmann (Other)
Responsible Party: Sponsor-Investigator, PD Dr. med. Eckart Bertelmann, Senior Consultant, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA1/171/14
Record Dates: First submitted 2015-12-14; First posted 2015-12-17 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Cataract
Keywords: Multifocal Intraocular Lens; Binocular Trifocality; Cataract Surgery; Spectacle Independence; Intermediate Vision; Photopic Vision; Mesopic Vision; Scotopic Vision; Binocular Vision
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Binocular cataract surgery with phacoemulsification and implantation of multifocal intraocular lenses — Binocular implantation of the combination of AMO® Tecnis® multifocal intraocular lenses with an addition of +2.75 D in the distance-dominant eye and +3.25 D in the fellow eye.
  Other Names: AMO® Tecnis® multifocal intraocular lenses with an addition of +2.75 D (ZKB00) and +3.25 D (ZLB00) are used.

SUMMARY:
The objective of this study is to assess the visual outcome after the combined binocular implantation of +2.75 D and +3.25 D full-diffractive multifocal intraocular lenses.

DETAILED DESCRIPTION:
Bifocal multifocal intraocular lenses (MIOL) are effective in achieving good uncorrected visual acuities in the distance and the near. However, the intermediate vision is of increasing relevance for everyday's life. Several multifocal intraocular lenses have been developed to improvement intermediate vision. Nonetheless, those systems still possess adverse photic effects and do not garantuee spectacle independence. Therefore, the combination of a lower-addition bifocal intraocular lense in the distance-dominant eye with a higher-addition bifocal intraocular lense in the fellow-eye might be a promising approach to address these drawbacks of current binocular and trifocal intraocular lenses.

ELIGIBILITY:
Inclusion Criteria:

* clinically significant cataract
* endothelial cell count: patients aged 18-75 years: > 1000 cells/mm2; patients > 75 years: > 750 cells/mm2
* absence of vision-limiting corneal or retinal comorbidities
* capability to understand the informed consent

Exclusion Criteria:

* expected postoperative astigmatism > 0.75 diopters
* irregular astigmatism
* dilated pupil diameter < 3 mm
* corneal and fundus abnormalities that might cause visual impairments
* inability to attend follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Visual acuities in the far, intermediate and near | 1 month
  Visual acuities are tested under photopic conditions at 5 m, intermediate (80 cm) and patient-preferred near distance (≈ 40 cm).
Visual acuities in the far, intermediate and near | 3 months
  Visual acuities are tested under photopic conditions at 5 m, intermediate (80 cm) and patient-preferred near distance (≈ 40 cm).
Mesopic vision | 1 month
  Mesopic visual acuities are tested under high-contrast, low-contrast and low-contrast with glare.
Mesopic vision | 3 months
  Mesopic visual acuities are tested under high-contrast, low-contrast and low-contrast with glare.
Scotopic contrast sensitivity | 1 month
  Scotopic contrast sensitivity are tested at 0.1 cd/m2, 0.032 cd/m2 and 0.1 cd/m2 with glare.
Scotopic contrast sensitivity | 3 months
  Scotopic contrast sensitivity are tested at 0.1 cd/m2, 0.032 cd/m2 and 0.1 cd/m2 with glare.

SECONDARY OUTCOMES:
Spectacle independence in the far, intermediate and near | 3 months
  Spectacle independence as stated by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Eckart Bertelmann, MD, Principal Investigator — Charité - University Medicine Berlin, Department of Ophthalmology
Locations (1):
- Charité - University Medicine Berlin, Department of Ophthalmology, Berlin, Germany

REFERENCES:
- [Background] Kretz FT, Koss MJ, Auffarth GU; ZLB00 Study Group. Intermediate and near visual acuity of an aspheric, bifocal, diffractive multifocal intraocular lens with +3.25 D near addition. J Refract Surg. 2015 May;31(5):295-9. doi: 10.3928/1081597X-20150423-02. PMID 25974967
- [Background] Kretz FT, Gerl M, Gerl R, Muller M, Auffarth GU; ZKB00 Study Group. Clinical evaluation of a new pupil independent diffractive multifocal intraocular lens with a +2.75 D near addition: a European multicentre study. Br J Ophthalmol. 2015 Dec;99(12):1655-9. doi: 10.1136/bjophthalmol-2015-306811. Epub 2015 May 18. PMID 25987651
- [Background] Vega F, Alba-Bueno F, Millan MS, Varon C, Gil MA, Buil JA. Halo and Through-Focus Performance of Four Diffractive Multifocal Intraocular Lenses. Invest Ophthalmol Vis Sci. 2015 Jun;56(6):3967-75. doi: 10.1167/iovs.15-16600. PMID 26098463
- [Background] Vega F, Millan MS, Vila-Terricabras N, Alba-Bueno F. Visible Versus Near-Infrared Optical Performance of Diffractive Multifocal Intraocular Lenses. Invest Ophthalmol Vis Sci. 2015 Nov;56(12):7345-51. doi: 10.1167/iovs.15-17664. PMID 26562168
- [Background] Kim JS, Jung JW, Lee JM, Seo KY, Kim EK, Kim TI. Clinical Outcomes Following Implantation of Diffractive Multifocal Intraocular Lenses With Varying Add Powers. Am J Ophthalmol. 2015 Oct;160(4):702-9.e1. doi: 10.1016/j.ajo.2015.07.021. Epub 2015 Jul 21. PMID 26209232